CLINICAL TRIAL: NCT03759483
Title: Diagnostic Efficacy of Convolutional Neural Network Based Algorithm in Differentiation of Glaucomatous Visual Field From Non-glaucomatous Visual Field
Brief Title: Diagnostic Efficacy of CNN in Differentiation of Visual Field
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center，Director of Institution of Drug Clinical Trials, Sun Yat-sen University
Other Study IDs: 2018KYPJ125
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diagnositic Efficacy of Deep Convolutional Neural Network in Differentiation of Glaucoma Visual Field From Non-glaucoma Visual Field
Keywords: Deep convolutional neural network; Visual field; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI group: The visual field reports in this group will be evaluated by the convolutional neural network.
  Interventions: Diagnostic Test: AI diagnostic algorithm
- Human group: The visual field reports in this group will be evaluated by 3 ophthalmologists independently.

INTERVENTIONS:
Diagnostic Test: AI diagnostic algorithm — The visual fields collected would be assessed by the algorithm and ophthalmologists independently. The performance of the algorithm and the ophthalmologists would be compared, including accuracy, AUC, sensitivity and specificity.
  Other Names: Standard diagnostic procedure
  Groups: AI group

SUMMARY:
Glaucoma is currently the leading cause of irreversible blindness in the world. The multi-center study is designed to evaluate the efficacy of the convolutional neural network based algorithm in differentiation of glaucomatous from non-glaucomatous visual field, and to assess its utility in the real world.

DETAILED DESCRIPTION:
Glaucoma is the world's leading cause of irreversible blind, characterized by progressive retinal nerve fiber layer thinning and visual field defects. Visual field test is one of the gold standards for diagnosis and evaluation of progression of glaucoma. However, there is no universally accepted standard for the interpretation of visual field results, which is subjective and requires a large amount of experience. At present, artificial intelligence has achieved the accuracy comparable to human physicians in the interpretation of medical imaging of many different diseases. Previously, we have trained a deep convolutional neural network to read the visual field reports, which has even higher diagnostic efficacy than ophthalmologists. The current multi-center study is designed to evaluate the efficacy of the convolutional neural network based algorithm in differentiation of glaucomatous from non-glaucomatous visual field, compare its performance with ophthalmologists and to assess its utility in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18;
2. Informed consent obtained;
3. Diagnosed with specific ocular diseases;
4. Able to perform visual field test

Exclusion Criteria:

Incomplete clinical data to support diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from clinics in different eye centers across China. Each subject must be diagnosed based on comprehensive medical tests and medical records. The leading center will read all the medical data to give out diagnosis as the gold standard.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
AUC value of convolutional neural network in differentiation of Glaucoma visual field from non-glaucoma visual field | from Jan 2019 to Jan 2020

SECONDARY OUTCOMES:
Sensitivity and specificity of convolutional neural network in detection of glaucoma visual field | from Jan 2019 to Jan 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No